CLINICAL TRIAL: NCT01314391
Title: Pilot Case-Control Study of WT1 Mutations in Wilms Tumor Patients Who Develop ESRD
Brief Title: Biomarkers in Blood and Tumor Tissue Samples From Patients With Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN11B1; COG-AREN11B1 (Other: Children's Oncology Group); NCI-2011-02850 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN11B1 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Cancer; Renal Failure
Keywords: stage I Wilms tumor; stage II Wilms tumor; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; renal failure
MeSH Terms: conditions — Kidney Neoplasms; Renal Insufficiency; Wilms Tumor | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and Tumor tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in blood and tumor tissue samples from patients with Wilms tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether Wilms Tumor (WT) patients without WT1-associated congenital anomalies or syndromes, but with end-stage renal disease (ESRD) unrelated to progressive bilateral tumors, carry germline WT1 mutations.
* To determine whether non-syndromic WT1 germline mutation carriers have a substantially higher incidence of ESRD than do WT patients who do not harbor WT1 mutations.

OUTLINE: Archived blood and tumor tissue specimens (or DNA isolated from these samples) are analyzed for WT1 mutations by gene sequencing and PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Wilms Tumor (WT)
* Patients who participated in the NWTS-5 protocol

  * Non-syndromic patients who developed end-stage renal disease (ESRD) during 5-10 years for reasons other than progressive bilateral WT
  * Matched control patients who had not developed ESRD by the time (since WT onset) of ESRD diagnosis
* Blood and tumor tissue samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Diagnosis of Wilms Tumor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Higher incidence of ESRD in non-syndromic WT patients with germline WT1 mutations than WT patients without WT1 mutations

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Huff, PhD, Principal Investigator — M.D. Anderson Cancer Center